CLINICAL TRIAL: NCT06763640
Title: Prognostic Value of Deep Learning-Derived Tumor-Infiltrating Lymphocyte Percentage in Nasopharyngeal Carcinoma: a Prospective Observational Study
Brief Title: Prognostic Value of TIL in Nasopharyngeal Carcinoma
Status: Enrolling by invitation | Type: Observational
Sponsor: Jiangxi Provincial Cancer Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SKJP1320241975
Record Dates: First submitted 2024-12-25; First posted 2025-01-08 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Nasopharyngeal Carcinoma (NPC)
Keywords: nasopharyngeal carcinoma; digital pathology images; deep learning; tumor-infiltrating lymphocytes; metastatic risk
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Our center plans to conduct a prospective, multicenter, observational study aimed at observing the percentage of TIL infiltration calculated using deep learning methods based on digital pathological images, and analyzing its prognostic significance in nasopharyngeal carcinoma, in order to help guide personalized treatment.

ELIGIBILITY:
Inclusion Criteria：

* Histopathology confirms nasopharyngeal carcinoma;
* At the initial treatment, there was no evidence of distant metastasis, and the staging was II-III (AJCC 9th);
* Age range of 18-70 years old, KPS ≥ 80 points;
* Having good organ function; The following conditions must be met: Hematology: White blood cell count>3.0 × 109/L; Absolute neutrophil count (ANC)>1.5 × 109/L; Hb>90g/L； Platelets>100 × 109/L; Albumin ≥ 3g/dL Liver function: Bilirubin ≤ 1.5 times the upper limit of normal (ULN), AST and ALT ≤ 3 times ULN, and alkaline phosphatase (ALP) ≤ 3 times ULN • International normalized ratio (INR) or prothrombin time (PT) or activated partial thromboplastin time (APTT) ≤ 1.5 times ULN; • Renal function: Serum creatinine ≤ 1.5 times ULN or creatinine clearance rate ≥ 60mL/min.
* Patients who are willing and able to comply with visit arrangements, treatment plans, laboratory tests, and other research procedures;
* Willing to comply with arrangements during the research period and cannot participate in any other clinical studies related to drugs and medical devices;
* Patients sign a formal informed consent form to indicate that they understand that this study complies with hospital policies.
* Sufficient tissue stored in wax blocks suitable for scientific research use.

Exclusion Criteria:

* Merge with other malignant tumors
* Individuals with a history of severe immediate hypersensitivity to any medication used in this study
* No capacity for civil conduct or limited capacity for civil conduct;
* Abuse of drugs or alcohol addiction, patients with physical or mental illnesses, and those deemed by the researchers to have a complete or thorough understanding of the possible complications of this study;
* Other serious acute or chronic medical conditions (including immune-mediated colitis, inflammatory bowel disease, non-infectious pneumonia, pulmonary fibrosis) or mental illnesses (including dementia and epilepsy, recent, past year, or active suicidal ideation or behavior) that may increase the risks associated with the study protocol treatment, or may interfere with the interpretation of study results and (based on the researcher's judgment) make patients unsuitable for participation in this study, or laboratory test abnormalities;
* Previously diagnosed with immunodeficiency or known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS) related diseases;
* Pregnant or lactating female patients, male or female patients who have fertility but are unwilling or unable to use contraception for at least one year throughout the study period and after the end of the treatment plan.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Jiangxi Cancer Hospital
Sampling Method: Non-Probability Sample
Enrollment: 216 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease Free Survival (DFS) | 3 Years
  DFS was defined as the interval from the date of diagnosis to the data of disease recurrence or death

SECONDARY OUTCOMES:
Overall Survival | 3 Years
  Overall Survival was defined as the interval from the date of diagnosis to the date of death for any cause
Distant Metastasis-free Survival | 3 Years
  DMFS was defined as the interval from the date of diagnosis to the data of distant metastases or censored at the date of last follow-up
Locoregional Recurrenc-free Survival | 3 Years
  LRRFS was defined as the interval from the date of diagnosis to the data of locoregional recurrence or censored at the date of last follow-up
Objective Response Rate | During induction chemotherapy (up to 3 months)
  Objective response rate is defined as the proportion of patients with a complete response or partial response to treatment according to Response Evaluation Criteria in Solid Tumors (RECIST1.1)

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangxi Cancer Hospital, Nanchang, Jiangxi, China